CLINICAL TRIAL: NCT03099122
Title: A Prospective, Multi-center, Single-arm, Interventional Study of Thymoglobuline® Induction Therapy in Adult Recipients of Donated After Cardiac Death Kidney Transplant in China
Brief Title: A Study of Thymoglobuline® Induction Therapy in Adult Recipients of Donated After Cardiac Death Kidney Transplant
Acronym: START-DCD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: THYMOL07282; U1111-1178-5402 (Other: UTN)
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: End-stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Antilymphocyte Serum; Tacrolimus; Methylprednisolone; Mycophenolic Acid; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Thymoglobuline (Experimental): A cumulative dose of Thymoglobuline will be given intravenously, with a variable interval dose. Methylprednisolone will be given as induction therapy, according to institutional practice.
  Tacrolimus, mycophenolate, and prednisone will be given as maintenance therapies.
  Interventions: Biological: Rabbit Anti-thymocyte Immunoglobulin; Drug: Tacrolimus; Drug: Methylprednisolone; Drug: Mycophenolate mofetil; Drug: Mycophenolate Na; Drug: prednisone

INTERVENTIONS:
Biological: Rabbit Anti-thymocyte Immunoglobulin — Pharmaceutical form: creamy-white powder
  Route of administration: intravenous
  Other Names: Thymoglobuline
Drug: Tacrolimus — Pharmaceutical form: tablet
  Route of administration: oral
Drug: Methylprednisolone — Pharmaceutical form: powder
  Route of administration: intravenous
Drug: Mycophenolate mofetil — Pharmaceutical form: capsule
  Route of administration: oral
Drug: Mycophenolate Na — Pharmaceutical form: capsule
  Route of administration: oral
Drug: prednisone — Pharmaceutical form: tablet
  Route of administration: oral

SUMMARY:
Primary Objective:

To investigate the efficacy of the standard dose of Thymoglobuline® induction therapy for preventing acute rejection (AR) after transplantation among recipients of Donated after Cardiac Death (DCD) kidney transplant.

Secondary Objectives:

* To evaluate delayed graft function (DGF), graft and patient survival after kidney transplant.
* To evaluate adverse events of Thymoglobuline® throughout the study.
* To explore possible risk factors of AR and DGF in patients with DCD kidney transplant.
* To evaluate AR and DGF under different risk stratifications and explore an description optimal induction therapy regimen for recipients of DCD kidney transplant.

DETAILED DESCRIPTION:
The total study duration per patient is 6.5 months.

ELIGIBILITY:
Inclusion criteria :

* Male or female.
* Patient is a Chinese recipient of kidney transplant for the first time.
* Patient is a recipient of kidney allograft from Chinese donors donated after cardiac death (including kidney donated after brain death followed by circulatory death).
* Recipient's age is between 18 to 65 years old (including 18 years).
* Donor's age is more than 5 years old.
* Recipient's weight is greater than or equal to 50 kg but less than or equal to 80 kg.
* Patient fully understands the study and signs the informed consent form (ICF) prior to any study procedure.

Exclusion criteria:

* Patient is a multiple organ transplant recipient.
* Recipient with previous kidney or other organ transplant history.
* Recipient and donor have incompatible blood types.
* Recipient and donor have 5 or 6 mismatched human leucocyte antigen (HLA).
* Recipient is known to have an active infection or active chronic infection, or is seropositive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV Ab), or human immunodeficiency virus (HIV). (Serological test results within 12 months before transplantation are acceptable.)
* Recipient with cytomegalovirus (CMV) immunoglobulin G (IgG) negative who receives an allograft from CMV IgG positive donor (CMV IgG [D+/R-]).
* Any systemic infection requiring continuous treatment at enrolment, but prophylactic treatment of CMV and/or Pneumocystis carinii pneumonia (PCP) is allowed.
* Recipient has severe thrombocytopenia or leucopenia before operation (platelet count <75,000/ul, or the number of white blood cells <3,000 cells/mm3).
* Serum levels of alanine aminotransferase (ALT), aspartate aminotransferase (AST) or gamma glutamine transferase (GGT) ≥3ULN (upper limit of normal) within 1 week before transplantation, and not normalized at time of transplantation.
* Recipient has a history of malignancy within 5 years.
* Recipient with history of allergy and anaphylaxes to rabbit proteins or to any excipients.
* Recipient has known contraindications to the administration of Thymoglobuline®.
* Recipient has taken other investigational drugs or prohibited therapy for this study within 1 month or 5 of half-lives from screening, whichever is longer.
* Recipient has previously used Thymoglobuline®, or has participated in any clinical trial of any other medicine or device within 30 days before signing ICF.
* Pregnant or lactating women.
* Male and female patients do not agree to practice medically acceptable contraception (i.e., barrier or pharmacologic: male patient must use condoms or his female partner must take oral contraceptives; the male partner of a female patient must use condoms ) for at least 6 months following the study treatment.
* Conditions/situations such as:

  * Recipient not suitable for participation, whatever the reason, as judged by the Investigator, including medical, clinical, or psychosocial conditions, or patient potentially at risk of noncompliance to study procedures.
  * Donor known or suspected to have active infection before donation (such as blood cultures positive, seropositive for hepatitis B surface antigen [HBsAg], or antibody against hepatitis C virus [HCVAb], or human immunodeficiency virus [HIV]) or hypersensitive recipients (eg, panel reactive antibody [PRA] positive) before transplantation, judged by the Investigator.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with biopsy-proven acute rejection events | 6 months

SECONDARY OUTCOMES:
Percentage of delayed graft function events | 6 months
Duration of delayed graft function events | 6 months
Percentage of survived grafts | 6 months
Percentage of survived patients | 6 months
Assessment of acute rejection risk factors | 6 months
Assessment of delayed graft function risk factors | 6 months
Percentage of acute rejection events in different risk stratifications | 6 months
Percentage of delayed graft function events in different risk stratifications | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- CHINA, China, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org